CLINICAL TRIAL: NCT02099279
Title: Prognostic Value Cardiac Dysfunction Assessed by Bedside Echocardiography in Critically Ill COPD Patients Requiring Mechanical Ventilation
Status: Completed | Type: Observational
Sponsor: Jinhua Central Hospital (Other)
Responsible Party: Principal Investigator, Zhongheng Zhang, intensivist, Jinhua Central Hospital
Other Study IDs: echo_COPD; echo and COPD (Registry Identifier: echo and COPD)
Record Dates: First submitted 2014-03-23; First posted 2014-03-28 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2014-03

CONDITIONS: COPD Patients; Mechanical Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- echocardiography examination
  Interventions: Device: echocardiography examination

INTERVENTIONS:
Device: echocardiography examination — patients underwent echocardiography examination

SUMMARY:
Chronic obstructive lung disease (COPD) is a major cause of morbidity and mortality, and is a major reason for ICU admission. Cardiac function is often impaired in this disease but its association with clinical outcome has not been fully established. The study aims to investigate the association between cardiac dysfunction and clinclial outcomes.

DETAILED DESCRIPTION:
This is a prospective observational study conducted in a 47-bed mixed ICU of tertiary academic teaching hospital. The study will be performed between January 2014 to December 2015. All patients meeting the diagnostic criteria of AECOPD and admitted to ICU are potentially eligible for the present study. Relevant demographics and laboratory measurements are obtained. Transthoracic echocardiography (TTE) is performed immediately after ICU admission by experienced intensivists. Cox proportional hazard regression model is fitted by using stepwise forward selection and backward elimination technique. If linear assumption is not satisfied, the linear spline function will be used.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients experiencing episode of exacerbation and require mechanical ventilation were admitted to ICU

Exclusion Criteria:

* COPD patients admitted to ICU due to other reasons (major surgery, ischemic heart disease, and renal failure)
* moribund and expected to die within 48 hours
* with Do-Not-Resuscitation order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients meeting the diagnostic criteria of AECOPD and admitted to ICU are potentially eligible for the present study. The diagnosis of AECOPD is based on that defined in Global Initiative for Chronic Obstructive Pulmonary Disease. AECOPD is defined using definitive criteria with at least two of the following major symptoms: increased dyspnea, increased sputum purulence, increased sputum volume; or one major and one minor symptom: nasal discharge/congestion, wheeze, sore throat and cough for at least two consecutive days.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
28-day mortality | 28 days after ICU admission
  28 days after ICU admission; if a patient leave ICU before 28-days, it is considered as censored.

SECONDARY OUTCOMES:
duration of mechanical ventilation | from ICU admission to extubation, an expected average of 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Chen Kun, MB, Study Chair — Jinhua Municipal Central Hospital
Locations (1):
- Jinhua municipal central hospital, Jinhua, Zhejiang, China

REFERENCES:
- [Derived] Zhang Z, Chen L, Chen K, Ni H. The prognostic value of cardiac dysfunction assessed by bedside echocardiography in critically ill patients with COPD requiring mechanical ventilation: a study protocol. BMJ Open. 2014 Sep 25;4(9):e005359. doi: 10.1136/bmjopen-2014-005359. PMID 25256186